CLINICAL TRIAL: NCT01884103
Title: Field Triage of Older Adults Who Experience Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Manish Shah, Associate Professor of Emergency Medicine, Public Health Sciences, and Geriatrics, University of Rochester
Other Study IDs: 1U01CE002175 (NIH)
Record Dates: First submitted 2013-06-13; First posted 2013-06-21 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Traumatic Brain Injury; TBI
Keywords: TBI; Trauma; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EMS Providers: Field Triage Decision-making for older adult patients with potential TBI.

SUMMARY:
Our overall goal in this proposed study is to describe the current prehospital trauma triage process for older adult (age≥55) patients with suspected Traumatic Brain Injury (TBI), to identify the effect of certain medications (anticoagulants and platelet inhibitors) on TBI-related need for trauma center services, and to identify novel TBI screening strategies that are feasible for use in the prehospital setting.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is major source of disability and death for older adults. Of particular concern is that older adults most frequently sustain TBIs after low-mechanism injuries, such as falls from standing height, and frequently use anticoagulants and platelet inhibitors, which place them at risk for worse clinical outcomes. With the growth of the older adult population and the expanding use of anticoagulants and platelet inhibitors, TBI among older adults will continue to be a major source of morbidity and mortality unless methods are identified to improve outcomes in this unique population.

Building upon our long-standing and highly successful EMS research laboratory that has specifically focused on the triage of injured patients and the prehospital care of older patients and employing a combination of qualitative and quantitative methods, we will collect data from a large, multi-county catchment area that includes multiple EMS agencies, urban and rural environments, as well as trauma centers and non-trauma centers. In this study, we will: 1) identify candidate neurologic scales to maximize detection of high-risk older adult TBI patients; 2) characterize the current trauma triage process used by EMS providers to identify older patients with suspected TBI and patients taking anticoagulants and/or platelet inhibitors; 3) assess the public health burden of TBI among older adult EMS patients taking anticoagulants and/or platelet inhibitors; 4) assess the predictive ability of novel prehospital-based neurologic screening strategies to identify high-risk older adult TBI patients in the prehospital setting who require TBI-related trauma center care. Findings from this study have the potential to shift clinical practice in the prehospital setting by informing future recommendations for the identification of TBI among older adults taking anticoagulants or platelet inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* EMS Provider arriving with a patient who is injured >=55 years old

Exclusion Criteria:

* No systematic exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency Medical Service (EMS) providers who transport injured older adult patients to any of the participating Emergency Departments in Rochester, NY.
Sampling Method: Non-Probability Sample
Enrollment: 4533 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of older adult EMS patients taking anticoagulants and/or platelet inhibitors who require TBI-related trauma center care. | Within 72 hrs of initiating EMS care
Sensitivity, specificity and overall classification accuracy of selected neurologic scales (including GCS, and a newly developed scale) used in the prehospital setting to maximize detection of high-risk older TBI patients. | Within 72 hrs of initiating EMS care

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, MD, MPH, Principal Investigator — University of Rochester